CLINICAL TRIAL: NCT02205060
Title: Interventionnal and Randomized Study Measuring Virtual Reality Cue Exposure for the Relapse Prevention of Tobacco Consumption Versus Cognitive and Behavioral Approaches Therapy
Brief Title: Virtual Reality Cue Exposurefor the Relapse Prevention of Tobacco Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013-A01253-42
Record Dates: First submitted 2014-07-25; First posted 2014-07-31 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Chronic Tabagism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- virtual reality exposure therapy (VRET) (Experimental)
  Interventions: Other: virtual reality exposure treatment
- cognitive and behavioral approaches therapy without VRET (Experimental)
  Interventions: Other: cognitive and behavioral approaches therapy

INTERVENTIONS:
Other: virtual reality exposure treatment
  Arms: virtual reality exposure therapy (VRET)
Other: cognitive and behavioral approaches therapy
  Arms: cognitive and behavioral approaches therapy without VRET

SUMMARY:
The therapeutic efficacy of virtual reality has been validated for the treatment of various mental disorders ,smoking behavior is the first preventable cause of death in developed countries However, after a successful withdrawal, a high relapse rate (between 40 and 70%)has been observed, which emphasize the urgent need to implement new strategies. Virtual reality cue exposure for the relapse of tobacco consumption

DETAILED DESCRIPTION:
Smoking behavior is the first preventable cause of death in developed countries (World.Health.Organisation, 2009).It is reinforced by the nicotine found in cigarettes. This compound is responsible for a notable dependence effect. As a result of mass consumption, this subsequent addiction of tobacco is a psychiatric disorder that represents a significant public health issue. In France, the latest health survey INEPS (2010) retrieved an increase of daily smokers with a prevalence of 28.7% among adults over 15 years (Beck et al., 2010). However, after a successful withdrawal, a high relapse rate (between 40 and 70%) (Hatsukami et al., 2008) has been observed, which emphasize the urgent need to implement new strategies. These relapses are due to the presence of conditions associated with tobacco consumption (drinking in bars or restaurant, coffee break at the workplace, etc.). (Garcia-Rodriguez et al., 2012). These same situations are difficult to reconstruct in the framework of a hospital or an office.

Virtual reality has been introduced in the field of psychiatry as a method entitled virtual reality exposure therapy (VRET). Virtual reality allows patients to interact with a virtual environment (Riva and Wiederhold, 2002). This media can therefore help to generate synthetic environments which represent risk situations for the patient in the context of relapse prevention.

The therapeutic efficacy of virtual reality has been validated for the treatment of various mental disorders (phobias, agoraphobia and post-traumatic stress, etc.) (Powers and Emmelkamp, 2008). These studies have shown that VRET was at least as effective as traditional CBT while providing immersive and controllable virtual environments. During the recent years, its scope has expanded to tobacco addiction (Garcia-Rodriguez et al., 2012), although this area of research remains in experimental field and requires carrying out ad-hoc clinical trials. Indeed, compared to the standard treatment, VRET offers various advantages for cue exposure, such as controlled environments and complex, dynamic interactive three-dimensional situations (virtual Bars, office and artificial smokers computerized restaurants, etc.). It features the possibility of gradually exposing the patient to situations considered to be of a "high risk of relapse" in the confidentiality of an office and repeating these procedures as often as necessary. Lastly it allows the therapist to guide the patient in real time helping them to modify emotions and addiction related cognitions.

ELIGIBILITY:
Inclusion Criteria:

* Smoking withdrawal for at least 1 week
* Age more than 18 years

Exclusion Criteria:

* Epilepsy
* Psychiatic desease
* Dementia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-08-05 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
evaluate the abstinence of tobacco consumption | 12 months
  The primary outcome measure is represented by the efficiency which will be defined in success / failure. The success is estimated at 6 months, from the abstinence of the patient. The abstinence is defined by the total absence of tobacco consumption

SECONDARY OUTCOMES:
assess the impact of this treatment strategy on depression | 12 months
  depression wil be assess by Beck Depression Inventory - BDI scale

OTHER OUTCOMES:
assess the impact of this treatment strategy on quality of life | 12 months
  quality of life will be assess by SF 12 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eric Malbos, MD, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Giovancarli C, Malbos E, Baumstarck K, Parola N, Pelissier MF, Lancon C, Auquier P, Boyer L. Virtual reality cue exposure for the relapse prevention of tobacco consumption: a study protocol for a randomized controlled trial. Trials. 2016 Feb 19;17:96. doi: 10.1186/s13063-016-1224-5. PMID 26892001